CLINICAL TRIAL: NCT01258153
Title: Double-blind, Randomised, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Oral Administration of Nepadutant in Infant Colic
Brief Title: Preliminary Efficacy and Safety Study of Oral Nepadutant in Infant Colic
Acronym: no-cry
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIC-03
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Infantile Colic
Keywords: Infantile Colic; tachykinin antagonist; Nepadutant
MeSH Terms: conditions — Colic | interventions — MEN 11420

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nepadutant Low Dose (Experimental)
  Interventions: Drug: Nepadutant oral solution
- Nepadutant High Dose (Experimental)
  Interventions: Drug: Nepadutant oral solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching Nepadutant oral solution

INTERVENTIONS:
Drug: Nepadutant oral solution — Oral administration once daily for 7 days
  Arms: Nepadutant Low Dose
Drug: Nepadutant oral solution — Oral administration once daily for 7 days
  Arms: Nepadutant High Dose
Drug: Placebo matching Nepadutant oral solution — Oral administration once daily for 7 days
  Arms: Placebo

SUMMARY:
This phase IIa study is designed as a multi-centre, multinational, randomised, double-blind, placebo controlled study in three parallel groups, with the aim to evaluate the efficacy and safety of Nepadutant given at two oral doses once daily for seven days in comparison to placebo in the treatment of infantile colic.

DETAILED DESCRIPTION:
Infant colic is a functional gastrointestinal disorders which affects up to the 30% of the infant population; it is primarily characterised by excessive inconsolable crying starting without any apparent cause and lasting for several hours per day.

Current non pharmacological interventions (e.g. message, restriction in maternal diet in breast-feeding infants) and pharmacological treatments (simethicone, antimuscarinic drugs) are largely unsatisfactory.

In animal models, Nepadutant reverse the exaggerated intestinal motility and sensitivity, induced by different stimuli, without producing inhibitory effects on these functions at baseline, suggesting that Nepadutant could have a therapeutic effect with no interference on physiological gastrointestinal transit.

This phase IIa study is designed to evaluate the efficacy of Nepadutant paediatric oral solution given once daily at two doses in comparison to placebo.

The experimental clinical phase encompasses the following periods:

* Screening period (no study medication) to be done 7 to 4 days prior to randomisation
* Treatment period, lasting seven days with once daily administration
* Post treatment period, lasting seven days A safety follow-up visit will be performed approximately 1 month after the first administered dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants with diagnosis of infant colic according to the following modified Wessel criterion "paroxysm of irritability, fussing or crying that start and stop without obvious cause for >3h/day, >3 days/week for one week"
* Age > 4 weeks and < 20 weeks
* Infants breast-fed mixed fed or formula fed with a stable dietary regimen
* Normal growth
* History of no adequate response to conventional treatment alternatives which make the infants in need of medical treatment
* Willingness to refrain from use of antimuscarinic drugs, simethicone, dimethicone or antiacids during the study period.

Exclusion Criteria:

* Clinical evidence of allergies or other diseases which may cause crying and/or fussiness or may interfere with absorption or clearance of the drug.
* Suspect of gastroesophageal reflux disease (GERD)
* Suspect of cow milk allergy.

Ages: 4 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Koletzko, MD, Study Chair — Dr. v. Haunersches Kinderspital Ludwig Maximilians University D- 80337 München, Germany
Locations (8):
- Dr. von Haunersches Kinderspital Ludwig Maximilians Universität München, München, Germany
- Klinika Patologii Noworodkow, Niemowlat I Kardiologii, Dzieciecy Szpital Kliniczny, Lublin, Poland
- Russia (5):
  - Federal Scientific Clinical Center of Children Hematology, Oncology and Immunology, Moscow
  - Moscow State Healthcare Institution Municipal Pediatric health center № 10, Moscow
  - Moscow State Medical University, Moscow
  - St. Petersburg State Pediatric Medical Academy, Saint Petersburg
  - St. Petersburg State Institution of Healthcare Municipal Pediatric health center № 35, Saint Petersburg
- Pediatrics Department of Clinical sciences Umeå university, Umeå, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Nepadutant Low Dose: Nepadutant oral solution 0.1mg/kg: Oral administration once daily for 7 days
- Nepadutant High Dose: Nepadutant oral solution 0.5mg/kg: Oral administration once daily for 7 days
Period: Overall Study
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Started | 40 | 38 | 37
Completed | 39 | 37 | 36
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 113 : ITT - defined as the safety population randomised with at least 24h diary recording post 1st dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 36 | 113
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 11.03 (4.909) | 11.34 (5.147) | 10.92 (4.686) | 11.1 (4.881)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 17 | 51
  Male | 18 | 25 | 19 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 38 | 37 | 36 | 111
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 5.22 (1.129) | 5.24 (1.267) | 5.61 (1.419) | 5.35 (1.275)
Feeding Mode [Number; unit: participants] — Feeding mode: 1 data missing in high dose - 0.5mg/kg (37 subjects instead of 38)
  participants
    Breast Fed | 27 | 29 | 29 | 85
    Formula Fed | 9 | 7 | 7 | 23
    Mixed Fed | 3 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change of the Mean Daily Crying and Fussing Time for Three Consecutive Days While on Treatment Versus Baseline.
Description: Efficacy assessment to be measured through "baby's day" diary recorded for three consecutive days while on treatment (i.e. starting from 6 pm on Day 4 and continued for 72 hours) vs baseline (i.e. starting from 6 pm on Day -4 until 1st treatment administration).
Time Frame: Baseline and one week
Population: 112 instead of 113, because 1 subject had no records at baseline and therefore the outcome could not be measured
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Number analyzed (Participants) | 38 | 38 | 36
Minutes
  Baseline | 284.57 (89.298) | 273.6 (86.356) | 283.91 (80.201)
  End of Treatment | 185.8 (100.97) | 154.4 (102) | 192.7 (85.41)
  Change | -96.9 (74.12) | -119.2 (97.13) | -91.2 (76.2)

2. Secondary Outcome: Percentage of 'Responder' Babies at the End of Treatment Period.
Description: Response is defined as a decrease of at least 50% of crying and fussing time during the last 3 days on treatment vs baseline.
Time Frame: baseline and one week
Population: 112 instead of 113, because 1 subject had no records at baseline and therefore the outcome could not be measured
Measure: Number; unit: Responders Rate (% of responders babies)
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Number analyzed (Participants) | 38 | 38 | 36
Responders Rate (% of responders babies) | 36.8 | 55.3 | 19.4

3. Secondary Outcome: Absolute Change in the Overall Parental Judgment After the First Dose of Treatment Versus Baseline
Description: On a daily basis parents expressed an overall judgement on the study treatment effect based on a 6 rate categorical scale from 0 to 5 (where 0 is for "Not at all" and 5 is "Extremely".
  The question was "How frustrating to you was your baby's crying today?")
Time Frame: 1 day
Population: ITT - defined as the safety population randomised with at least 24h diary recording post 1st dose of study treatment
Measure: Mean (Standard Deviation); unit: Score range 0-5
Units Other Than Participants: Questionnaires completed by parents
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Number analyzed (Participants) | 39 | 38 | 36
Number analyzed (Questionnaires completed by parents) | 38 | 37 | 35
Score range 0-5 | -0.38 (0.771) | -0.68 (0.884) | -0.34 (0.596)

4. Secondary Outcome: Absolute Change in the Overall Parental Judgment at the End of Treatment Versus Baseline
Description: as for outcome 3
Time Frame: 1 week
Population: ITT - defined as the safety population randomised with at least 24h diary recording post 1st dose of study treatment
Measure: Mean (Standard Deviation); unit: Score range 0-5
Units Other Than Participants: Questionnaires completed by parents
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Number analyzed (Participants) | 39 | 38 | 36
Number analyzed (Questionnaires completed by parents) | 38 | 36 | 36
Score range 0-5 | -1.24 (0.909) | -1.75 (1.186) | -1.23 (1.044)

5. Secondary Outcome: Absolute Change in the Overall Parental Judgment After Treatment Discontinuation Versus Baseline
Description: as for outcome 3
Time Frame: 10 days
Population: ITT - defined as the safety population randomised with at least 24h diary recording post 1st dose of study treatment
Measure: Mean (Standard Deviation); unit: Score range 0-5
Units Other Than Participants: Questionnaires completed by parents
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Number analyzed (Participants) | 39 | 38 | 36
Number analyzed (Questionnaires completed by parents) | 38 | 37 | 36
Score range 0-5 | -1.35 (0.857) | -1.78 (1.176) | -1.39 (0.896)

6. Secondary Outcome: Safety and Tolerability Will be Assessed in Terms of Frequency and Severity of AEs as Well as Frequency of Clinically Significant Changes in Physical Examination and Lab Test.
Description: Safety and tolerability will be assessed for the Safety Population (all patients who received the study drug) in terms of frequency and severity of AEs as well as frequency of clinically significant changes in physical examination and lab test.
Time Frame: up to four weeks
Population: All patients receiving the study drug (114)
Measure: Number; unit: Adverse events
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Number analyzed (Participants) | 40 | 38 | 36
Adverse events | 9 | 6 | 5

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Nepadutant Low Dose | Nepadutant High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/38 | 0/36
Other Adverse Events (participants affected / at risk) | 9/40 | 6/38 | 5/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nepadutant Low Dose (N=40) | Nepadutant High Dose (N=38) | Placebo (N=36)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Hospitalization for Bronchitis in a 10 weeks-old male infant. The investigator considered the SAE as unlikely related to the study drug. It resolved without sequel.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nepadutant Low Dose (N=40) | Nepadutant High Dose (N=38) | Placebo (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Salivary ipersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 1 | 0
Gamma -GT abnormal (Investigations) | 1 | 0 | 0
Crying (Nervous system disorders) | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study cannot be submitted for presentation, abstract, poster exhibition, or publication by the investigator until Menarini Ricerche S.p.A. has reviewed/commented and agreed to any publication.